CLINICAL TRIAL: NCT02389699
Title: Comparison of the Efficacy of Intra-operative Radiation Therapy After Conserving Surgery With Post-operative Whole Breast Radiotherapy for Women With Ductal Carcinoma in Situ
Brief Title: Comparison of Intra-operative Radiotherapy With Post-operative Radiotherapy for Women With Ductal Carcinoma in Situ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liao Ning (Other)
Responsible Party: Sponsor-Investigator, Liao Ning, Guangdong Academy of Medical Sciences, Guangdong Academy of Medical Sciences
Organization: Guangdong Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGHBCRG-IORT-WRT-DCIS
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breast Neoplasms
Keywords: Intermediate and high grade ductal carcinoma in situ （DCIS）
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraoperative Radiotherapy (Experimental): Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  Interventions: Radiation: Intraoperative Radiotherapy
- whole breast radiation (Active Comparator): WRT:whole breast radiation after BCS with 46-50 Gy
  Interventions: Radiation: Whole breast radiation

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy — Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  Arms: Intraoperative Radiotherapy
Radiation: Whole breast radiation — whole breast radiation after BCS with 46-50 Gy
  Arms: whole breast radiation

SUMMARY:
Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation during surgery followed by external-beam radiation to the entire breast may kill more tumor cells.The clinical trial is conducting to compare the effectiveness of radiation therapy during surgery and whole-breast radiation therapy in treating women who have undergone breast-conversing surgery for Intermediate or high grade ductal carcinoma in situ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Tumor diameter < 5 cm
* Intermediate or high grade ductal carcinoma in situ
* Informed consent

Exclusion Criteria:

* No informed consent
* Tumor size > 3,5 cm
* Low grade ductal carcinoma in situ
* Invasive carcinoma
* No indication for a boost

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
ipsilateral breast tumor recurrence rate after surgery within five years | Within 5 years after surgery
  Within 5 years after surgery,we should evaluate ipsilateral breast tumor recurrence and Disease free survival as the most important outcome measure
Disease free survival after surgery within five years | Within 5 years after surgery
  Within 5 years after adjuvant chemotherapy,we should evaluateDisease free survival(DFS) rates as thet important outcome measure.

SECONDARY OUTCOMES:
Overall survival after surgery within ten years | Within ten years after surgery
  After surgery,we should evaluate overall survival (OR)rates as the secondary important outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Ning, MD,PhD, Study Director — Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China